CLINICAL TRIAL: NCT03296046
Title: Epidemiologic Study of Persistent Polyclonal B-cell Lymphocytosis (PPBL) - Observatory 1990-2012
Brief Title: Epidemiologic Study of Persistent Polyclonal B-cell Lymphocytosis (PPBL)
Acronym: LPLB
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/PSS/LPLB/LESESVE//MS
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Persistent Polyclonal B-Cell Lymphocytosis
MeSH Terms: conditions — Persistent Polyclonal B-Cell Lymphocytosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood (30 ml) taken during routine care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PPBL patients
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — 30 ml

SUMMARY:
The main purpose of this study is the description of all French cases of PPBL and the establishment of minimal criteria for the pathology diagnosis and its follow-up.

The secondary objective is the immunologic and genetic characterization of lymphoid cells causing the disease.

ELIGIBILITY:
Inclusion Criteria:

* PPBL diagnosis established during a previous medical visit

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PPBL patients in France
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-11-13 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Relevant medical history | Baseline
Complete blood count | Baseline
Administration of first-line treatment or not | Baseline

SECONDARY OUTCOMES:
Lymphocyte phenotype | Baseline

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - group GFHC and intergroup LLC (GCFLL-MW / GOELAMS), Marseille
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No